CLINICAL TRIAL: NCT00153647
Title: A Study to Assess the Success Rate of Cap-Assisted Colonoscopy Versus Regular Colonoscopy for the First or Repeated Colonoscopy (CAC Study)
Brief Title: A Study to Assess Cap-Assisted Colonoscopy Versus Regular Colonoscopy for the First or Repeated Colonoscopy
Acronym: CAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Francis K CHAN, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAC Study
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2007-08

CONDITIONS: Colonoscopy; Lower Gastrointestinal Tract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Cap-assisted Colonoscopy
  Interventions: Procedure: Cap-assisted colonoscopy
- 2 (Placebo Comparator): Regular Colonoscopy
  Interventions: Procedure: Cap-assisted colonoscopy

INTERVENTIONS:
Procedure: Cap-assisted colonoscopy — Cap-assisted colonoscopy
  Arms: 1
Procedure: Cap-assisted colonoscopy — Cap-assisted colonoscopy
  Arms: 2

SUMMARY:
The primary aim of the study is to increase the success rate of cecal intubation in first colonoscopy and in repeated colonoscopy for the first failed procedure. The secondary aims are to assess the procedure time, the terminal ileum intubation rate, the endoscopist satisfaction score, the patients' acceptance, the complication rate of these two procedures, and the intravenous sedative drugs used.

DETAILED DESCRIPTION:
Currently there is no consensus in how to improve the success rate of colonoscopy procedure given the fact that 10% of the procedures may fail. It has been suggested that using variable stiffness colonoscope (a colonoscope with a shaft that the stiffness can be altered), or even more sophisticated magnetic imaging colonoscopy (colonoscopy performed under a magnetic position detection sensor), could improve the success rate. However, these kinds of equipment are either expensive or not always available in the daily clinical practice. From some recent studies it was shown that adding a transparent cap to the tip of the colonoscope may improve the procedure success rate without increasing the complication rate of the procedure. The cost of the cap is cheap and it is available in almost every endoscopy center. Therefore the cap-assisted colonoscopy method may be an alternative which may improve the success rate of colonoscopy procedure, and reduce the pain and discomfort related to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo their first colonoscopy examination

Exclusion Criteria:

* Patients had received colonoscopy examination before
* Patients had prior colorectal surgery done (apart from appendectomy)
* Known to have colonic stricture or obstructing tumor from the results of other investigations such as CT scan or barium enema
* Presence of acute surgical conditions such as severe colitis, megacolon, ischemic colitis and active gastrointestinal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2005-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The success rate of cecal intubation | 24 hours

SECONDARY OUTCOMES:
The procedure time to achieve cecal intubation | 24 hours
Success rate in achieving terminal ileum intubation | 24 hours
The procedure time to achieve terminal ileum intubation | 24 hours
Complications related to the procedure | 24 hours
The procedure difficulty as assessed by the endoscopist using a 10 cm visual analog scale | 24 hours
The procedure difficulty of polypectomy if indicated as assessed by the endoscopist using a 10 cm visual analog scale | 24 hours
The patient's pain score as assessed by the patient using a visual analog scale right after he regains full consciousness, which is assessed by accurately performing a deduction test (100 minus 7 test, correct for three deductions), before discharge | 24 hours
The dose of the intravenous drugs used | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Y T Lee, MD, Principal Investigator — Department of Medicine & Therapeutics, Prince of Wales Hospital
Locations (2):
- China (2):
  - Endoscopy Center, Alice Ho Miu Ling Nethersole Hospital, Hong Kong
  - Endoscopy Center, Prince of Wales Hospital, Hong Kong